CLINICAL TRIAL: NCT05113056
Title: The Pulsed Field Ablation System Study for Atrial Fibrillation (PFA-AF)
Brief Title: AcQForce Pulsed Field Ablation-CE
Acronym: PFA-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acutus Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP-23
Record Dates: First submitted 2021-10-28; First posted 2021-11-09 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Atrial Arrhythmia; Atrial Fibrillation
Keywords: atrial fibrillation; ablation; pulsed field ablation (PFA)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: The patient population will consist of men and women between the ages of 18 - 80 years, presenting for a de novo ablation for atrial fibrillation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-randomized (Experimental): All subjects will be ablated using the Acutus Medical Pulsed Field Ablation System (PFA System) in the management of their atrial fibrillation.
  Interventions: Device: Acutus Medical Pulsed Field Ablation System

INTERVENTIONS:
Device: Acutus Medical Pulsed Field Ablation System — All subjects will be treated using the Acutus Medical Pulsed Field Ablation System (PFA System) to treat their atrial fibrillation.

SUMMARY:
The Pulsed Field Ablation System Study for Atrial Fibrillation (PFA-AF)

DETAILED DESCRIPTION:
This clinical study is designed to evaluate the safety and performance of the PFA System in the ablation treatment of atrial fibrillation (AF). Data will be used to support regulatory submissions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 18 to 80 years at time of consent
2. Clinically indicated and scheduled for a de novo catheter ablation of AF
3. Willing and able to provide written informed consent to participate in the study and agree to comply with all follow-up visits and evaluations for the duration of the study.

Exclusion Criteria:

1. In the opinion of the investigator, any contraindication to the planned atrial ablation, including anticoagulation contraindications, atrial thrombus, renal failure, or sepsis.
2. Continuous episodes of AF duration lasting longer than 12-months
3. Atrial arrhythmias secondary to electrolyte imbalance, thyroid disease, or any other reversible or non-cardiac cause.
4. Previous history of left atrial ablation (including surgical treatment) for AF/AT/AFL.
5. Structural heart disease or cardiac history as described below:

   1. Left ventricular ejection fraction (LVEF) < 35%
   2. Left atrial size > 60 mm
   3. Evidence of heart failure (NYHA Class III or IV)
   4. Unstable angina or ongoing myocardial ischemia
   5. Recent myocardial infarction
   6. Severe uncontrolled systemic hypertension
   7. Moderate or severe valvular heart disease (stenosis or regurgitation).
   8. Interatrial baffle, closure device, patch, or patent foramen ovale (PFO) occluder.

   l. Presence of a left atrial appendage occlusion device. j. Previous PV stenting or evidence of PV stenosis.
6. Body Mass Index (BMI) > 42 kg/m2
7. History of blood clotting or bleeding disease.
8. ANY prior history of documented cerebral infarct (stroke), or systemic embolism (excluding post-operative deep vein thrombosis (DVT)).
9. History of obstructive sleep apnea not currently being treated.
10. Pregnant or lactating (current or anticipated during study follow-up).
11. Any other condition that, in the judgment of the Investigator, makes the patient a poor candidate for this procedure, the study or compliance with the protocol (includes vulnerable patient population, mental illness, addictive disease, terminal illness with a life expectancy of less than two years, extensive travel away from the research center).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who are free from device/procedure related Major Adverse Events | 6 months
  The Primary Endpoint for Safety is an analysis of the proportion of subjects who are free from device/procedure related Major Adverse Events (MAEs) that occur following the ablation procedure through 6-months.
Acute documentation of pulmonary vein isolation (PVI) for each treated pulmonary vein (PV) | 20 minutes post ablation
  The Primary Endpoint for efficacy is the number of subjects where ablation of each accessible pulmonary vein (PV) resulted in confirmation of electrical isolation of the pulmonary vein (PVI) 20 minutes following the last index PFA/RF application with the investigational device

SECONDARY OUTCOMES:
Analysis of all identified SAEs, SADEs, and UADEs | 12 months
  The Secondary Endpoint for Safety is a recording and analysis of all identified serious adverse events (SAEs), serious adverse device effects (SADEs), and unanticipated adverse device effects (UADEs).
Subjects with freedom from an atrial arrhythmia | 12 months
  The Secondary Endpoint for Performance is documentation of subjects with freedom from an atrial arrhythmia at 12-months post index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Petr Neuzil, MD, Principal Investigator — Na Homolce Hospital
Locations (1):
- Na Homolce Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided